CLINICAL TRIAL: NCT05644522
Title: Power Forward Study: A Cross-Sector, Multisite Clinical Trial of a Powered Knee-Ankle-Foot Orthosis
Brief Title: Nomad P-KAFO Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STU00217395
Record Dates: First submitted 2022-11-28; First posted 2022-12-09 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cerebrovascular Accident; Post-polio Syndrome; Spinal Cord Injuries; Multiple Sclerosis; Muscular Dystrophy; Paralysis
MeSH Terms: conditions — Stroke; Postpoliomyelitis Syndrome; Spinal Cord Injuries; Multiple Sclerosis; Muscular Dystrophies; Paralysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A receives the intervention Nomad KAFO first; fitting & training will occur with the intervention and will then be used for a 3 month home trial, followed by outcomes testing. Group A then will cross over and train with their own Traditional Assistive Device and will then use their own device for a 3 month home trial, followed by outcomes testing.
  Interventions: Device: Indego Nomad® Powered Knee-Ankle-Foot Orthosis (P-KAFO) (Parker Hannifin Corp., Cleveland, OH)
- Group B (Active Comparator): Group B receives training in their own Traditional Assistive Device first; training will occur with their own Traditional Assistive Device and will then use their own device for a 3 month home trial, followed by outcomes testing. Group B then will cross over and receive the intervention Nomad KAFO; fitting & training will occur with the intervention and will then be used for a 3 month home trial, followed by outcomes testing.
  Interventions: Device: Indego Nomad® Powered Knee-Ankle-Foot Orthosis (P-KAFO) (Parker Hannifin Corp., Cleveland, OH)

INTERVENTIONS:
Device: Indego Nomad® Powered Knee-Ankle-Foot Orthosis (P-KAFO) (Parker Hannifin Corp., Cleveland, OH) — The Nomad is a microprocessor-controlled knee-ankle-foot orthosis P-KAFO that incorporates a motor for powered movement assistance and an electronic brake for stance support. The system provides active assistance for knee flexion and extension during the swing phase of gait, reliable stance phase locking at any knee angle, and reliable unlocking without requiring user-generated knee or hip extension torque.

SUMMARY:
The goal of this clinical trial is to evaluate the impact of using the Nomad powered KAFO in people who have had a musculoskeletal or neurological injury that has affected their ability to walk. The main questions it aims to answer are to quantify the effectiveness of the Nomad in improving mobility, balance, frequency of falls, and quality of life in individuals with lower-extremity impairments compared to their own brace, over three months of daily home and community use.

Participants will:

* Wear a sensor that records everyday activities and mobility.
* Perform measures of mobility and different activities of participation using their own brace.
* Perform measures of mobility and different activities of participation using the Nomad powered KAFO

ELIGIBILITY:
Inclusion Criteria:

* Regular and compliant use of a unilateral or bilateral KAFO or SCO or other passive KAFOs for impairment due to neurological or neuromuscular disease, orthopedic disease, or trauma
* Cognitive ability to understand and follow the study protocol; willingness to provide informed consent
* Willing to wear and charge an activity monitor for three-months home trials.

Exclusion Criteria:

* Flexion contracture in the knee and/or hip joint in excess of 15 degrees
* Non-correctable knee varus/valgus in excess of 15 degrees
* Severe spasticity
* Inability to stabilize the trunk with or without assistive devices (crutches, canes, etc.)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in 10 Meter Walk Test speed | Baseline, Post 3-month home trials with each device
  A test to measure the change of speed of both self selected and fastest walking speeds

SECONDARY OUTCOMES:
Six Minute Walk Test | Baseline, Post 3-month home trials with each device
  A test to measure how much distance is traveled over the course of 6 minutes.
Berg Balance Test | Baseline, Post 3-month home trials with each device
  A test of standing balance
Functional Gait Assessment | Baseline, Post 3-month home trials with each device
  A test of postural stability during walking tasks
Hill Assessment Index | Baseline, Post 3-month home trials with each device
  Used to assess different gait patterns during ascent or descent of slopes
Stair Assessment Index | Baseline, Post 3-month home trials with each device
  Used to assess functional abilities during ascent and descent of stairs
Timed Up and Go | Baseline, Post 3-month home trials with each device
  A functional mobility test to measure how long it takes to rise from a chair, walk 3 meters, turn around, and return back to a sitting position in the chair.
Activities Specific Balance Confidence Scale | Baseline, Post 3-month home trials with each device
  A self-report questionnaire designed to measure fear of falling across 16 items.
Modified Falls Efficacy Scale | Baseline, Post 3-month home trials with each device
  A self-report questionnaire designed to measure fear of falling across 14 items.
Orthotics and Prosthetics User Survey | Baseline, Post 3-month home trials with each device
  A self-report questionnaire designed to evaluate the outcome of orthotic and prosthetic services.
World Health Organization Quality of Life | Baseline, Post 3-month home trials with each device
  A self-report questionnaire that measures an individual's perceived quality of life.
EQ5D-5L | Baseline, Post 3-month home trials with each device
  A self-report questionnaire that measures quality of life with mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Numeric Pain Rating Scale | Baseline, Post 3-month home trials with each device, and as needed throughout course of study.
  A measure of perceived pain intensity
Borg Rate of Perceived Exertion | Baseline, Post 3-month home trials with each device, and as needed throughout course of study
  A measure of perceived exertion during an activity
Manual Muscle Test | Screening, Baseline, Post 3-month home trials with each device
  A rating of overall gross muscle strength
Range of Motion (both passive and active) | Screening, Baseline, Post 3-month home trials with each device
  A measurement of overall joint mobility of both lower extremities
Six Minute Push Test | Baseline, Post 3-month home trials with each device
  A test to determine distance traveled in a wheelchair with self-propulsion over the course of 6 minutes.

OTHER OUTCOMES:
Cross Walk Blinking Signal Test | Baseline, Post 3-month home trials with each device
  Measuring the time needed to cross a designated street
Community Mobility | During each 3 month home trial with each device.
  Measured by wearing an activity monitor to capture motion / step counts
Self Reported Goals | Baseline, Post 3-month home trials with each device
  Subjects will be interviewed to understand their self-reported functional goals.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States